CLINICAL TRIAL: NCT03747224
Title: A Phase 1 Single and Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamic Effects of ARO-ANG3 in Adult Healthy Volunteers and in Dyslipidemic Patients
Brief Title: Study of ARO-ANG3 in Healthy Volunteers and in Dyslipidemic Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AROANG1001
Record Dates: First submitted 2018-11-16; First posted 2018-11-20 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Dyslipidemias; Familial Hypercholesterolemia; Hypertriglyceridemia
MeSH Terms: conditions — Dyslipidemias; Hyperlipoproteinemia Type II; Hypertriglyceridemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ARO-ANG3 (Experimental)
  Interventions: Drug: ARO-ANG3
- Placebo (Placebo Comparator)
  Interventions: Drug: sterile normal saline (0.9% NaCl)

INTERVENTIONS:
Drug: ARO-ANG3 — single or multiple doses of ARO-ANG3 by subcutaneous (sc) injections
  Arms: ARO-ANG3
Drug: sterile normal saline (0.9% NaCl) — calculated volume to match active treatment
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetcs and pharmacodynamics of single- and multiple doses of ARO-ANG3 in healthy adult volunteers and in dyslipidemic patients including familial hypercholesterolemia and severe hypertriglyceridemia.

ELIGIBILITY:
Inclusion Criteria:

* Women of child bearing potential must have a negative pregnancy test, cannot be breastfeeding and must be willing to use contraception
* Willing to provide written informed consent and to comply with study requirements
* On a stable diet for at least 4 weeks with no plans to significantly alter diet or weight over course of study
* Normal electrocardiogram (ECG) at Screening

Exclusion Criteria:

* Clinically significant health concerns
* Regular use of alcohol within one month prior to Screening
* Use of an investigational agent or device within 30 days prior to dosing or current participation in an investigational study
* Recent use of illicit drugs
* Use of more than two tobacco/nicotine containing or cannabis products per month within 6 months prior to drug administration (applicable only to Normal Healthy Volunteers)

NOTE: additional inclusion/exclusion criteria may apply, per protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-05-17 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) Possibly or Probably Related to Treatment | Up to 113 (+/- 3 days) post-dose

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of ARO-ANG3: Maximum Observed Plasma Concentration (Cmax) | Single dose phase: Up to 48 hours post-dose
PK of ARO-ANG3: Time to Maximum Plasma Concentration (Tmax) | Single dose phase: Up to 48 hours post-dose
PK of ARO-ANG3: Terminal Elimination Half-Life (t1/2) | Single dose phase: Up to 48 hours post-dose
PK of ARO-ANG3: Area Under the Plasma Concentration Versus Time Curve From Zero to 24 Hours (AUC0-24) | Single dose phase: Up to 48 hours post-dose
PK of ARO-ANG3: Area Under the Plasma Concentration Versus Time Curve From Zero to infinity (AUCinf) | Single dose phase: Up to 48 hours post-dose
Reduction in Fasting Serum ANGPTL3 from Pre-Dose Baseline | Baseline, Up to Day 113 (+/- 3 days)

CONTACTS AND LOCATIONS:
Locations (6):
- Australia (3):
  - Research Site 2, Camperdown, New South Wales
  - Research Site 3, Adelaide, South Australia
  - Research Site 1, Nedlands
- New Zealand (3):
  - Research Site 4, Grafton, Auckland
  - Research Site 5, Papatoetoe, Aukland
  - Research Site 6, Christchurch

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Watts GF, Schwabe C, Scott R, Gladding PA, Sullivan D, Baker J, Clifton P, Hamilton J, Given B, Melquist S, Zhou R, Chang T, San Martin J, Gaudet D, Goldberg IJ, Knowles JW, Hegele RA, Ballantyne CM. RNA interference targeting ANGPTL3 for triglyceride and cholesterol lowering: phase 1 basket trial cohorts. Nat Med. 2023 Sep;29(9):2216-2223. doi: 10.1038/s41591-023-02494-2. Epub 2023 Aug 25. PMID 37626170
- [Derived] Ying Q, Chan DC, Watts GF. Angiopoietin-like protein 3 inhibitors and contemporary unmet needs in lipid management. Curr Opin Lipidol. 2021 Jun 1;32(3):210-212. doi: 10.1097/MOL.0000000000000747. No abstract available. PMID 33900278